CLINICAL TRIAL: NCT00668915
Title: Arthroplasty Rehabilitation Score - Can we Predict the Short Term Postoperative Outcome?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: rehabtjr-HMO-CTIL
Record Dates: First submitted 2008-04-28; First posted 2008-04-29 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Primary arthroplasty

SUMMARY:
Total joint arthroplasty are common operations among the elderly population. The postoperative patients' rehabilitation process may be influenced by a variety of factors, such as age, BMI, perioperative hemoglobin levels, pain perception, comorbidities, etc. Nevertheless, only a few well controlled studies evaluated the effect of various factors on patients' rehabilitation short-term outcome. Furthermore, no scale has been developed, that can predict patients' rehabilitation and functioning levels 6 weeks postoperatively. In the current study we wish to evaluate the effect on patients' function that the following factors have: age, BMI, admission and discharge hemoglobin levels, pain perception, type of operation (TKA versus THA), intensity of postoperative physiotherapy, involvement of other joints by the primary pathology, comorbidities, and self assessed health status.

In order to quantify patients' level of functioning, several tests will be used: hand grip strength, Timed up and go test (TUG) and Oxford knee and hip score. The factors that will be found statistically significantly associated with level of functioning, will be used in an attempt to develop a scale that will predict the level of functioning 6 weeks postoperatively.

Such a scale can allow preoperative identification of patients at high risk of postoperative low functioning levels and the application of a unique rehabilitation program, for only these patients, in order to optimize their functioning.

DETAILED DESCRIPTION:
This is a prospective, analytical, approximately 6 months long study.

Population:

Approximately a 100 patients, scheduled for an elective arthroplasty will be recruited for the study:

* Males and females above 18 years of age, speaking Hebrew, English or Russian, scheduled for an elective unilateral (one joint) primary total joint arthroplasty of hip or knee.
* Available for follow up 1.5-2 months after the surgery.
* Willing to participate in the study.

Inclusion criteria:

1. Patient above the age of 18 and eligible to provide informed consent.
2. Scheduled for elective unilateral (one joint), primary total joint arthroplasty of hip or knee.
3. Stepping with the operated leg is allowed after the surgery.

Exclusion criteria:

1. Patients unwilling to participate.
2. Patients with complications preventing regular rehabilitation, e.g. Myocardial Infarction, Pulmonary Embolism, Pneumonia, and infection or fracture of the joint.
3. Patients with any complication that prevents stepping with the operated leg.

Design:

1. Prior to the scheduled operation, the following data regarding the patient will be collected:

   * Gender, age, height, weight.
   * Comorbidities (using Katz Score).
   * Type of scheduled operation.
   * Involvement by the primary pathology of joints other than the one being operated (by patient questioning).
   * Hemoglobin level at admission.
   * Self assessed health status (by patient questioning).
   * Pain perception in the operated leg (using VAS Score).

   In addition, the following tests will be performed:
   * Evaluation of muscle strength using handgrip machine.
   * Evaluation of motor functioning level using the TUG test and the Oxford knee and hip score.
2. During the postoperative hospitalization period, hemoglobin and CRP levels will be checked, and the patients will be evaluated for complications.
3. In the follow up visit, the following data will be collected:

   * Complications after discharge from hospital.
   * Blood transfusions in this period.
   * Duration of time in rehabilitation program, and intensity of physiotherapy given.

During the visit, the following tests will be performed:

* Evaluation of muscle strength using handgrip machine.
* Evaluation of motor functioning level, similar to the one performed preoperatively, using the TUG test and the Oxford knee and hip score.

ELIGIBILITY:
Inclusion Criteria:

1. Patient above the age of 18 and eligible to provide informed consent.
2. Scheduled for elective unilateral (one joint), primary total joint arthroplasty of hip or knee.
3. Stepping with the operated leg is allowed after the surgery.

Exclusion Criteria:

1. Patients unwilling to participate.
2. Patients with complications preventing regular rehabilitation, e.g. Myocardial Infarction, Pulmonary Embolism, Pneumonia, and infection or fracture of the joint.
3. Patients with any complication that prevents stepping with the operated leg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary arthroplasty
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)

PRIMARY OUTCOMES:
Oxford hip and knee score
Grip strength
Timed up and go test

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel